CLINICAL TRIAL: NCT04160117
Title: Impact of Short-course Colchicine Versus Placebo After Pulmonary Vein Isolation (IMPROVE-PVI): a Pilot Study
Brief Title: Impact of Short-course Colchicine Versus Placebo After Pulmonary Vein Isolation (IMPROVE-PVI Pilot)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMPROVE-PVI pilot
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation; Recurrence
MeSH Terms: conditions — Atrial Fibrillation; Recurrence | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Colchicine 0.6 mg p.o. twice daily for 10 days after catheter ablation for atrial fibrillation
  Interventions: Drug: Colchicine 0.6 mg
- Control (Placebo Comparator): Matching placebo p.o. twice daily for 10 days after catheter ablation for atrial fibrillation
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Colchicine 0.6 mg — p.o. twice daily for 10 days after catheter ablation for atrial fibrillation
  Arms: Intervention
Drug: Matching placebo — p.o. twice daily for 10 days after catheter ablation for atrial fibrillation
  Arms: Control

SUMMARY:
Recurrence is a common problem after catheter ablation for atrial fibrillation, affecting at least one out of three patients. Inflammation due to the procedure may contribute to pulmonary vein reconnection and, thus, failure of catheter ablation.

This pilot study will assess whether a randomized, placebo-controlled, double-blind trial investigating a 10-day treatment with colchicine, a potent anti-inflammatory drug, to improve patient relevant outcomes after catheter ablation for atrial fibrillation is feasible.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Symptomatic atrial fibrillation and planned catheter-guided first or repeat ablation (pulmonary vein isolation) for atrial fibrillation (radiofrequency or cryoablation energy; concomitant ablation of the cavotricuspid isthmus and other lesions left at the discretion of the treating physician)
3. Written informed consent

Exclusion Criteria:

1. Ablation for left atrial tachycardia or isthmus-dependent atrial flutter only (i.e. without pulmonary vein isolation)
2. Administration of a strong inhibitor of CYP3A4 or p-gp (clarithromycin, erythromycin, telithromycin, cyclosporine, ketoconazole or itraconazole)
3. Known hypersensitivity to colchicine
4. Serious gastrointestinal disease (severe gastritis or diarrhea)
5. Clinically overt hepatic disease
6. Severe renal disease (eGFR< 30ml/min/1.73m2)
7. Clinically significant blood dyscrasia (e.g., myelodysplasia)
8. Absolute indication for or ongoing treatment with colchicine
9. Pregnant or breastfeeding women, or women of child-bearing potential who do not use a highly effective form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Average monthly enrollment rate | Through study completion (enrollment phase estimated to last 18 months, total study duration estimated to last 24 months)
  Average number of patients enrolled per month
Compliance with study treatment | From randomization until 10 days after catheter ablation
  Number of provided capsules taken (measured as a proportion of 20 capsules)
Rate of complete follow-up at 6 months | From inception until completion of the study
  This will describe the rate of patients for whom the 6-month follow visit can be completed

SECONDARY OUTCOMES:
Rate of non-infectious diarrhea | From randomization until 10 days after catheter ablation
  Three or more loose stools per day, in absence of an overt infectious cause
Rate of signs and symptoms of pericarditis | From randomization until 10 days after catheter ablation
  Evidence of new or worsening pericardial effusion on echocardiogram, friction rub on auscultation or pleuritic chest pain
Recurrence of atrial fibrillation within the first 2 weeks after catheter ablation | From randomization until 2 weeks after catheter ablation for atrial fibrillation
  Any episode of atrial fibrillation lasting > 30 seconds within 2 weeks after catheter ablation for atrial fibrillation. Atrial flutter or other forms of atrial tachycardia are included in this definition
Recurrence of atrial fibrillation between 10-15 weeks after catheter ablation | Between week 10 and 15 after catheter ablation for atrial fibrillation
  Any episode of atrial fibrillation lasting > 30 seconds between 10-15 weeks after catheter ablation for atrial fibrillation. Atrial flutter or other forms of atrial tachycardia are included in this definition
Rate of patients with composite clinical endpoint | Through study completion (estimated to be up to 24 months)
  Emergency department visit: Patient seeking medical attention at any emergency department or Hospitalization for cardiovascular cause: Minimum of one overnight stay in hospital for cardiovascular reason (e.g. recurrence of atrial fibrillation, atrial flutter, atrial tachycardia; hypotension; hypertension; heart failure; myocardial infarction; bleeding, stroke etc.) or Cardioversion: Pharmacological or electrical attempt of or restoring sinus rhythm, irrespective of success of the procedure or Repeat ablation for atrial fibrillation, atrial flutter or left atrial tachycardia: Catheter-guided pulmonary vein isolation, or ablation of cavotricuspid isthmus, or ablation for other left atrial tachycardia (e.g. macro-reentrant tachycardia, focal tachycardia) after the index procedure
Rate of all-cause mortality | Through study completion (estimated to be up to 24 months)
  This will describe the rate of all-cause mortality during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Benz, MD, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton Health Sciences Corporation - Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benz AP, Amit G, Connolly SJ, Singh J, Acosta-Velez JG, Conen D, Deif B, Divakaramenon S, McIntyre WF, Mtwesi V, Roberts JD, Wong JA, Zhao R, Healey JS; IMPROVE-PVI Investigators. Colchicine to Prevent Atrial Fibrillation Recurrence After Catheter Ablation: A Randomized, Placebo-Controlled Trial. Circ Arrhythm Electrophysiol. 2024 Jan;17(1):e01238. doi: 10.1161/CIRCEP.123.012387. Epub 2023 Dec 21. PMID 38126206